CLINICAL TRIAL: NCT02365207
Title: Evaluating Local and Regional Immune Responses to Intravesical BCG Administration to Patients With Invasive Bladder Cancer
Brief Title: Intravesical BCG Administration to Patients With Invasive Bladder Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor accrual of subjects and lack of funding
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-002
Record Dates: First submitted 2015-02-03; First posted 2015-02-18 (Estimated); Results first posted 2019-11-05 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2018-09

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BCG treatment of invasive bladder cancer (Experimental): Invasive bladder cancer treated with 3-6 weeks of intravesical BCG
  Interventions: Drug: BCG strain of Mycobacterium bovis

INTERVENTIONS:
Drug: BCG strain of Mycobacterium bovis — Invasive bladder cancer treated with 3-6 weeks of intravesical BCG
  Other Names: BCG

SUMMARY:
Patients with invasive bladder cancer will be given 3-6 treatments (based on treatment response) BCG intravesically followed by a cystectomy.

DETAILED DESCRIPTION:
Patients with muscle invasive (≥T1) bladder cancer will be given 3-6 treatments (based on treatment response) intravesical TICE® BCG. BCG is an attenuated, live culture preparation of the Bacillus of Calmette and Guerin (BCG) strain of Mycobacterium bovis.

After completion of BCG treatments the patient will undergo a cystectomy. A portion of bladder tumor tissue and lymph nodes will be collected for research purposes during the cystectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Have suspected or known invasive (≥T1) bladder cancer
2. Be able to give informed consent
3. Be age 18 or older
4. Not be in an immunosuppressed state (e.g. HIV+, use of chronic steroids >1 month)

Exclusion Criteria:

1. Have non-invasive (<T1) bladder cancer
2. Unable to give informed consent
3. < 18 or older
4. Is in an immunosuppressed state (e.g. HIV+, use of chronic steroids >1 month)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-11; Primary Completion 2018-09-30 (Actual); Study Completion 2019-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Svatek, MD, Principal Investigator — University of Texas
Locations (1):
- MARC - The University of Texas Health Science Center, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BCG Treatment of Invasive Bladder Cancer
Started | 6
Completed | 4
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | BCG Treatment of Invasive Bladder Cancer
Number analyzed (Participants) | 6
Age, Customized [Mean (Full Range); unit: Years] | 63.5 [51 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 3
  White-non Hispanic | 3
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Ability of BCG to Enhance Tumor Specific Immunity
Description: The tumor specific immunity is measured by the change in T cell proliferation post-treatment compared to the pre-treatment assessment, which will require a sample size of at least 10
Time Frame: At cystectomy at 3-6 weeks after BCG treatment
Population: Data were not analyzed, since the study closed prematurely due to poor accrual and lack of funding. Since the change in T-cell proliferation required a sample size of at least 10 and only 4 subjects who were randomized completed. No data were analyzed for this study, since that sample size was not achieved.
Arm/Group | BCG Treatment of Invasive Bladder Cancer
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected during BCG administration at 3-6 weeks prior to cystectomy. Adverse events are only reported in the 5 subjects who received study drug.
Arm/Group | BCG Treatment of Invasive Bladder Cancer
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 3/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BCG Treatment of Invasive Bladder Cancer (N=5)
Abdominal fluid collection (Surgical and medical procedures) | 2 (2) — Unanticipated: Subject was hospitalized with symptoms unrelated to study intervention: Abdominal fluid collection, body ache, chills, leg pain and surgical wound skin dehiscence
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Unanticipated: unrelated to study intervention (subject hospitalized post surgery)
Acute renal failure (Renal and urinary disorders) | 1 (1) — Unanticipated: related to surgical procedure, not study intervention
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BCG Treatment of Invasive Bladder Cancer (N=5)
Gross hematuria (Renal and urinary disorders) | 2 (2)
Exploratory laparotomy (Blood and lymphatic system disorders) | 1 (1) — Unanticipated: unrelated to study drug: diagnosis of anemia prompted an exploratory laparotomy
Dysuria (Renal and urinary disorders) | 1 (4) — Painful and frequent urination which resolved within 24 hours
Abdominal cramps (Gastrointestinal disorders) | 1 (1) — Abdominal cramps
Nausea (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-23): https://cdn.clinicaltrials.gov/large-docs/07/NCT02365207/Prot_SAP_000.pdf